CLINICAL TRIAL: NCT07051122
Title: Personalised Nutrition for the Preterm Infant
Acronym: Pinpoint
Status: Completed | Type: Observational
Sponsor: University College Cork (Other)
Responsible Party: Principal Investigator, Mairead Kiely PhD, Professor, University College Cork
Other Study IDs: Pinpoint
Record Dates: First submitted 2025-06-19; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Preterm Infant Nutrition
Keywords: Nutrition; nutrient; preterm infant nutrition; preterm
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Preterm infants: * Gestational age <34 weeks
  * Birth weight ≤1800g

SUMMARY:
The aim of the Pinpoint observational study is to collect nutrition and health data in a cohort of preterm, low birth weight infants to investigate if their nutrition support is adequate. Results will inform nutritional requirements and monitoring of preterm infants for macronutrients and micronutrients.

DETAILED DESCRIPTION:
Background The goal of neonatal nutrition in the preterm infant is to achieve postnatal growth and body composition approximating that of a normal fetus of the same postmenstrual age and to obtain a functional outcome comparable to infants born at term. While international consensus guidelines for the nutritional management of preterm infants have been formulated, gaps between these nutrition guidelines and clinical practice have been extensively reported, resulting in nutritional deficits and inadequate growth and development.

A previous study of preterm infants (NCT01881256), showed that despite best practice guidelines, infants did not receive sufficient energy and protein to meet recommendations, which contributed to early growth failure. While some recent progress has been made in the field, with studies demonstrating reductions in cumulative nutrient deficits and improvements in growth after the optimisation of nutritional protocols, uncertainties still remain as to the nutritional requirements of preterm infants and how best to meet them. The nutritional management of preterm infants is complicated by their complex nutritional needs and different sources of nutrients as they progress through the neonatal course.

Challenge A major drawback is the lack of real-time feedback data on actual daily nutrient intakes of infants in the neonatal unit. Without this precise information, nutritional management is based on estimates, which can lead to nutritional deficits. The consequences of missed opportunities for optimal nutrient delivery may be far-reaching, in terms of inadequate growth and suboptimal developmental outcomes. Enhanced nutritional data collection and monitoring at the infant's cot-side in the neonatal unit would support more effective clinical decision-making, resulting in improved outcomes for infants.

Objective To collect extensive data on nutrition and health in preterm, low birth weight infants to inform development of bespoke software to track nutrient delivery in the neonatal unit. To describe relationships between nutrient delivery and nutritional status of iron and vitamin D and to analyse the impact of revised nutritional recommendations on nutrition and growth.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age <34 weeks
* Birth weight ≤1800g
* Parents/legally authorised representative provides signed and dated informed proxy consent within 48 hours of infant's birth.

Exclusion Criteria:

• Infants born with life-threatening congenital or chromosomal abnormalities.

Max Age: 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm infants born less than 34 weeks of gestation and under 1800 g birth weight
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Nutrient delivery | From enrolment up to 10 weeks
  Total energy, macronutrient and micronutrient delivery from all sources, including parenteral and enteral nutrition and nutritional supplements will be collected and analysed in MC Excel and our bespoke preterm nutrition software to calculate individual energy, macronutrient and micronutrient intakes (on a daily basis) for comparison with historical data and international recommendations.

SECONDARY OUTCOMES:
Infant weight | From enrolment to 6 months corrected age
  Infant weight in grammes
Infant length | From enrolment to 6 months corrected age
  supine length in centimetres

OTHER OUTCOMES:
Nutritional status of vitamin D | From enrolment for 10 weeks
  Laboratory analysis of microsamples of serum for markers of vitamin D metabolism (25(OH)D in nmol/L)
Nutritional status of iron | From enrolment to 10 weeks
  Laboratory analysis of serum ferritin (microg/L)
Body Composition | From enrolment to 6 months corrected age
  Fat mass and fat free mass by air displacement plethysmography in grammes
Electroencephalogram (EEG) | From enrolment to 6 months corrected age
  Quantitative Electroencephalogram (EEG) features recorded during sleep divided into four groups: EEG magnitude, spectral distribution, continuity, and connectivity.
Neurological development | From enrolment to 6 months corrected age
  Griffiths Scales of Child Development, Third Edition analysis of overall general development (GD) and five neurodevelopmental areas: foundations of learning (A), language and communication (B), eye and hand coordination (C), personal-social-emotional (D), and gross motor abilities (E), with lower scores indicating more severe developmental delay.

CONTACTS AND LOCATIONS:
Locations (1):
- Cork University Maternity Hospital, Infant Research Centre, University College Cork, Cork, Ireland

IPD SHARING:
Plan to Share IPD: No
These data were collected in a vulnerable and heterogenous population. The consent provided by parents did not include data sharing.